CLINICAL TRIAL: NCT00929435
Title: The Incidence of Methicillin Resistant Staphylococcus Aureus (MRSA) Nasal Carriage Among Resident Physicians
Brief Title: Incidence of Methicillin Resistant Staphylococcus Aureus (MRSA) Carriage Rates in Resident Physicians
Status: Terminated | Type: Observational
Why Stopped: Minimal enrollment
Sponsor: University of Oklahoma (Other)
Responsible Party: Principal Investigator, Gary Kinasewitz, Principal Investigator, University of Oklahoma
Other Study IDs: 14684
Record Dates: First submitted 2009-06-24; First posted 2009-06-29 (Estimated); Last update posted 2012-04-09 (Estimated); Status verified 2012-04

CONDITIONS: MRSA Colonization
Keywords: MRSA; Contact isolation; Incidence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- MRSA surveillance: Newly recruited resident physicians will be monitored for a year with nasal swabs monthly.

SUMMARY:
One hundred new residents will be recruited prior to the start of residency and followed prospectively for a year. Monthly nasal swabs will be performed to identify colonization with methicillin resistant staphylococcus aureus (MRSA).The proportion of study subjects colonized with MRSA at the end of 1 year will be calculated.

DETAILED DESCRIPTION:
This is a prospective observational study looking at the incidence of MRSA colonization. New residents will be monitored every month with nasal swabs.We would like to elucidate factors responsible for MRSA colonization in healthcare workers.We would like to see if health care workers who are colonized spontaneously cleared MRSA and if there was any factors involved.

Nasal swabs will be plated on the spot by trained individuals and the plates then incubated for 48 hours. Plates will be read by microbiologist after incubation.

ELIGIBILITY:
Inclusion Criteria:

* Study subjects will be newly appointed residents at the OU medical center

Exclusion Criteria:

* Previous MRSA infection
* Current use of mupirocin

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All newly recruited residents will be eligible for enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2009-06; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
To detect an increase in MRSA nasal carriage rate among newly appointed residents after 1 year of regular patient contact. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Gary T Kinasewitz, MD, Principal Investigator — University of Oklahoma
Locations (1):
- Oklahoma University health science center, Oklahoma City, Oklahoma, United States